CLINICAL TRIAL: NCT03949959
Title: Effectiveness of Conservative Multimodal Physiotherapy in Chronic Whiplash-associated Disorders With Facet-mediated Pain Undergoing Platelet Rich Plasma (PRP) Treatment: a Series of Single Case Experimental Designs (SCEDs).
Brief Title: Effectiveness of Physiotherapy Following PRP for Chronic Whiplash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: REB18-0724
Record Dates: First submitted 2019-04-11; First posted 2019-05-14 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Whiplash Injuries; Neck Injuries; Platelet Rich Plasma
Keywords: Physiotherapy
MeSH Terms: conditions — Whiplash Injuries; Neck Injuries

STUDY DESIGN:
Intervention Model Description: A Single Case Experimental Design (SCED) will be used to evaluate the intervention. Participants act as their own controls, and thus are exposed to both the treatment and control conditions. The study will be conducted and reported according to the Singe Case Reporting guidelines in BEhavioural Interventions (SCRIBE). A randomised, concurrent, multiple-baseline A1 (baseline control) - B (intervention)-A2 (follow-up withdrawal) design will be used to meet the methodological recommendations for SCEDs. Participants will be randomly allocated to a 5, 8 or 11 day baseline period during which they will undertake their usual activities. The baseline phase will be followed by a 6-week intervention period during which participants will participate in 10, one hour sessions with an experienced post-graduate trained physiotherapist. The intervention phase will be followed by a 12-week follow-up phase where participants will have no contact with the intervention personnel.
Who Masked: Participant
Masking Description: Participant is not made aware of intervention arm - treat as usual or physiotherapy. Radiologist providing PRP tells participant to refrain from treatment for 6-weeks, or to immediately commence physiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy (PRPt) (Experimental): The 6-week exercise program (2 sessions in each of weeks 1-4 and 1 session in each of weeks 5 and 6) will comprise specific individually-tailored exercises to improve the movement and control of the neck and shoulder girdle. The exercises will be of a low load nature and designed to be pain free. At the same time, the physiotherapist will provide pragmatic multimodal physiotherapy to facilitate ability to pursue exercises and guide the participant's return to normal activities. This specific treatment program has been described in detail (Jull et al., 2008; Ritchie et al., 2015b) and focuses on activating and improving the coordination and endurance capacity of the neck flexor, extensor and scapular muscles in specific exercises and functional tasks. Participants will also perform the exercises at home, once per day. Written and illustrated exercise instructions will be provided. The exercise program follows Australian guidelines for the management of chronic whiplash (TRACsa, 2008).
  Interventions: Other: Multimodal physiotherapy
- Wait and See (PRPu) (No Intervention): Individuals randomized to usual care will be provided with an advice booklet Whiplash Injury Recovery: A Self Help Guide (MAIC, Qld, 2nd edition). It provides information about whiplash; assurance about prognosis; advice to stay active and resume working as well as information on correct posture; pictorial descriptions of specific exercises for the neck and upper limbs and information on resuming functional daily activities. The booklet is based on the recommendations of the current Australian Guidelines for Whiplash Management (SIRA, 2014).
  Usual care involves a 'wait and see' approach (in combination with provision of home exercises) and will include weekly review appointments with a medical doctor, primarily to review the information in the booklet and progress the 'general' exercises and activity recommendations within the booklet. No hands-on physiotherapy will be provided. Education regarding PRP and associated healing cycles will also be provided during this time period.

INTERVENTIONS:
Other: Multimodal physiotherapy — Participants will undertake their usual activities for the 5, 8 or 11 day baseline period following PRP. Participants will begin the 6 week intervention period following this period during which time they will participate in 10 sessions with an experienced postgraduate physiotherapist. After these 6-weeks, participants will have no contact with intervention personnel during the 6-week follow-up period.
  Arms: Physiotherapy (PRPt)

SUMMARY:
The investigators will explore a standardized and previously published evidence-based conservative multimodal physiotherapy treatment fulfilling clinical practice guidelines in individuals with chronic whiplash-associated disorders (WAD) with facet-mediated pain (appropriate response to dual medial branch blocks) undergoing cervical facet joint Plasma-Rich Platelet (PRPt) and compare health outcomes to individuals' undergoing cervical facet joint PRP with usual care (PRPu), which consists of advice, supervised home exercise and pharmacological management for treatment of residual pain. To be clear, the investigators are not investigating the efficacy or effectiveness of cervical facet joint PRP - these individuals have already consented to proceed with PRP treatment. The investigators are evaluating the role of adjuvant conservative multimodal physiotherapy treatment. It must be noted that these patients have previously failed to respond to conservative physiotherapy. The investigators will use a design which is quite novel in physiotherapy, Single Case Experimental Designs (SCEDs). In contrast to an experimental group design in which one group is compared with another, participants in single-subject research provide their own control data for the purpose of comparison in a within-subject rather than a between-subjects design. SCEDs provide a method to determine response and benefit for every individual patient.

Therefore, the investigators will assess effectiveness of conservative multimodal physiotherapy for chronic WAD with facet-mediated pain undergoing cervical facet joint PRP, using patients as their own control, in a multiple baseline design.

DETAILED DESCRIPTION:
This will be a single case with randomized multiple baseline experimental design with enrolment of 3 patients undergoing PRPt, and 3 patients undergoing PRPu following PRP. There will be a variable length baseline (A1) and then a staggered start to provide internal validity - one patient starting at 5 days (post-PRP), one at 8 (post-PRP) and one at 11 days post-PRP, randomly allocated. This study will utilise an A1-B-A2 design: a baseline (A1 no intervention); intervention phase (B); and a no intervention (A2 follow up).

Primary outcome measures will be collected daily during this time period. The baseline phase will be followed by a 6-week intervention period (B). Participants will have 10 one hour sessions over a 6-week period. The intervention will be delivered by an experienced physiotherapist with postgraduate qualifications. During the intervention period, once or twice per week the daily collection of the primary outcome measures will coincide with the delivery of each intervention session. The intervention phase will be followed by a 12-week follow-up phase (A2) where participants will have no contact with the intervention personnel. This follow-up phase is implemented in order to determine the possible duration of improvement post intervention. All outcome measures will be collected at the completion of this 12-week follow-up period.

Secondary outcome measures for generalisation purposes will be collected prior to commencing PRP, at the end of the intervention period (which coincides with the commencement of the no-intervention period), and at the end of the no-intervention period; totalling 3 sampling points throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Grade II Whiplash Associated Disorder with > 80% relief of familiar neck pain after dual medial branch blocks
* > 12 weeks since injury and failed to respond to previous (> 6 weeks) conservative treatment
* Neck pain on numerical pain rating scale ≥ 4/10
* Neck Disability Index > 28%

Exclusion Criteria:

* Presence of dizziness symptoms
* Known or suspected serious spinal pathology (e.g. metastatic disease of the spine);
* Confirmed fracture or dislocation at time of injury (i.e., WAD Grade IV)
* Nerve root compromise (i.e., WAD Grade III)
* Spinal surgery in the past 12 months; and
* History of any mental health conditions such as bipolar disorder, psychosis, schizophrenia, anxiety, PTSD or severe depression
* Inability to stop taking anti-inflammatory medications for 3-days prior to, or 10-days following PRP
* Unable to understand +/- complete validated questionnaire items in English

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Pain, Enjoyment of Life and General Activity (PEG) | 12 weeks
  PEG measures average neck pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G) on the continuous numeric rating scale (NRS) of 0 to 10 during the last 24 hours (Krebs et al., 2009).
Self-efficacy whilst performing daily activities in chronic WAD. | 12 weeks
  This question will ask participants to identify "how confident are you in your ability to perform your daily tasks in the presence of your neck pain or disability?" with 1 indicating not at all confident; 2 indicating a little confident 3 indicating moderately confident; 4 very confident and 5 indicating extremely confident.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Up to 11 days + 12 weeks
  The NDI is a reliable and responsive measure of neck pain related disability, validated for use with individuals following whiplash injury (Vernon & Mior, 1991). The 10-item questionnaire includes activities of daily living that may be affected by neck pain. A percentage score will be calculated from the 0-5 Likert scored response to each question.
Patient Global Impression of Change (-3 to +3 scale) | Up to 11 days + 12 weeks
  This is a 7 point scale that requires the clinician to assess how much the patient's condition has improved or worsened relative to a baseline state at the beginning of the intervention. +/- 3 relates to Very Much Improved/Worse; +/- 2 to Much Improved/Worse; +/-1 Minimally Improved/Worse
Depression & Anxiety Stress Scales (DASS-21) | Up to 11 days + 12 weeks
  The DASS-21 consists of 21 questions, each reflecting a negative emotional symptom. It consists of 3 subscales: Depressive, Anxiety and Stress symptoms. Each question is Likert scored (0-3). The sum of the relevant 7 items for each subscale constitute the participants' scores for each subscale (Lovibond & Lovibond, 1995).
The Pain Catastrophizing Scale (PCS) | Up to 11 days + 12 weeks
  This scale is a 13-item scale to evaluate catastrophic thinking about pain. It is Likert scored (1-4).
Medical Outcomes Survey Short Form (SF-12) | Up to 11 days + 12 weeks
  This survey measures health related quality of life. The SF-12 contains 12 questions relating to the domains physical functioning; role limitations because of physical health problems; bodily pain; general health perceptions; vitality (energy/fatigue); social functioning; role limitations because of emotional problems; and general mental health (psychological distress and psychological well-being). Physical and mental component summary scores are computed using the 12 questions and range from 0 (lowest level of health) to 100 (highest level of health) (Ware et al, 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Smith, PhD, Principal Investigator — University of Calgary
Locations (1):
- Vivo Cura Health, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll LJ, Holm LW, Hogg-Johnson S, Cote P, Cassidy JD, Haldeman S, Nordin M, Hurwitz EL, Carragee EJ, van der Velde G, Peloso PM, Guzman J; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Course and prognostic factors for neck pain in whiplash-associated disorders (WAD): results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S83-92. doi: 10.1097/BRS.0b013e3181643eb8. PMID 18204405
- [Background] Curatolo M, Bogduk N, Ivancic PC, McLean SA, Siegmund GP, Winkelstein BA. The role of tissue damage in whiplash-associated disorders: discussion paper 1. Spine (Phila Pa 1976). 2011 Dec 1;36(25 Suppl):S309-15. doi: 10.1097/BRS.0b013e318238842a. PMID 22020601
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Jull G, Sterling M, Kenardy J, Beller E. Does the presence of sensory hypersensitivity influence outcomes of physical rehabilitation for chronic whiplash?--A preliminary RCT. Pain. 2007 May;129(1-2):28-34. doi: 10.1016/j.pain.2006.09.030. Epub 2007 Jan 10. PMID 17218057
- [Background] Kaneoka K, Ono K, Inami S, Hayashi K. Motion analysis of cervical vertebrae during whiplash loading. Spine (Phila Pa 1976). 1999 Apr 15;24(8):763-9; discussion 770. doi: 10.1097/00007632-199904150-00006. PMID 10222526
- [Background] Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch SM, Kroenke K. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. J Gen Intern Med. 2009 Jun;24(6):733-8. doi: 10.1007/s11606-009-0981-1. Epub 2009 May 6. PMID 19418100
- [Background] Lamb SE, Gates S, Williams MA, Williamson EM, Mt-Isa S, Withers EJ, Castelnuovo E, Smith J, Ashby D, Cooke MW, Petrou S, Underwood MR; Managing Injuries of the Neck Trial (MINT) Study Team. Emergency department treatments and physiotherapy for acute whiplash: a pragmatic, two-step, randomised controlled trial. Lancet. 2013 Feb 16;381(9866):546-56. doi: 10.1016/S0140-6736(12)61304-X. Epub 2012 Dec 19. PMID 23260167
- [Background] Lillie EO, Patay B, Diamant J, Issell B, Topol EJ, Schork NJ. The n-of-1 clinical trial: the ultimate strategy for individualizing medicine? Per Med. 2011 Mar;8(2):161-173. doi: 10.2217/pme.11.7. PMID 21695041
- [Background] Lord SM, Barnsley L, Wallis BJ, Bogduk N. Chronic cervical zygapophysial joint pain after whiplash. A placebo-controlled prevalence study. Spine (Phila Pa 1976). 1996 Aug 1;21(15):1737-44; discussion 1744-5. doi: 10.1097/00007632-199608010-00005. PMID 8855458
- [Background] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Background] McDonald GJ, Lord SM, Bogduk N. Long-term follow-up of patients treated with cervical radiofrequency neurotomy for chronic neck pain. Neurosurgery. 1999 Jul;45(1):61-7; discussion 67-8. doi: 10.1097/00006123-199907000-00015. PMID 10414567
- [Background] Michaleff ZA, Maher CG, Lin CW, Rebbeck T, Jull G, Latimer J, Connelly L, Sterling M. Comprehensive physiotherapy exercise programme or advice for chronic whiplash (PROMISE): a pragmatic randomised controlled trial. Lancet. 2014 Jul 12;384(9938):133-41. doi: 10.1016/S0140-6736(14)60457-8. Epub 2014 Apr 4. PMID 24703832
- [Background] Nguyen RT, Borg-Stein J, McInnis K. Applications of platelet-rich plasma in musculoskeletal and sports medicine: an evidence-based approach. PM R. 2011 Mar;3(3):226-50. doi: 10.1016/j.pmrj.2010.11.007. PMID 21402369
- [Background] Quinn KP, Winkelstein BA. Detection of altered collagen fiber alignment in the cervical facet capsule after whiplash-like joint retraction. Ann Biomed Eng. 2011 Aug;39(8):2163-73. doi: 10.1007/s10439-011-0316-3. Epub 2011 May 3. PMID 21538155
- [Background] Ritchie C, Hendrikz J, Jull G, Elliott J, Sterling M. External validation of a clinical prediction rule to predict full recovery and ongoing moderate/severe disability following acute whiplash injury. J Orthop Sports Phys Ther. 2015 Apr;45(4):242-50. doi: 10.2519/jospt.2015.5642. PMID 25827122
- [Background] Ritchie C, Hendrikz J, Kenardy J, Sterling M. Derivation of a clinical prediction rule to identify both chronic moderate/severe disability and full recovery following whiplash injury. Pain. 2013 Oct;154(10):2198-2206. doi: 10.1016/j.pain.2013.07.001. Epub 2013 Jul 4. PMID 23831865
- [Background] Romeiser Logan L, Hickman RR, Harris SR, Heriza CB. Single-subject research design: recommendations for levels of evidence and quality rating. Dev Med Child Neurol. 2008 Feb;50(2):99-103. doi: 10.1111/j.1469-8749.2007.02005.x. PMID 18201299
- [Background] Sampson S, Gerhardt M, Mandelbaum B. Platelet rich plasma injection grafts for musculoskeletal injuries: a review. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):165-74. doi: 10.1007/s12178-008-9032-5. PMID 19468902
- [Background] Siegmund GP, Myers BS, Davis MB, Bohnet HF, Winkelstein BA. Mechanical evidence of cervical facet capsule injury during whiplash: a cadaveric study using combined shear, compression, and extension loading. Spine (Phila Pa 1976). 2001 Oct 1;26(19):2095-101. doi: 10.1097/00007632-200110010-00010. PMID 11698885
- [Background] Smith AD, Jull G, Schneider G, Frizzell B, Hooper RA, Dunne-Proctor R, Sterling M. Cervical radiofrequency neurotomy reduces psychological features in individuals with chronic whiplash symptoms. Pain Physician. 2014 May-Jun;17(3):265-74. PMID 24850108
- [Background] Smith AD, Jull G, Schneider GM, Frizzell B, Hooper RA, Sterling M. Modulation of Cervical Facet Joint Nociception and Pain Attenuates Physical and Psychological Features of Chronic Whiplash: A Prospective Study. PM R. 2015 Sep;7(9):913-921. doi: 10.1016/j.pmrj.2015.03.014. Epub 2015 Mar 21. PMID 25805617
- [Background] Smith AD, Jull G, Schneider G, Frizzell B, Hooper RA, Sterling M. A comparison of physical and psychological features of responders and non-responders to cervical facet blocks in chronic whiplash. BMC Musculoskelet Disord. 2013 Nov 4;14:313. doi: 10.1186/1471-2474-14-313. PMID 24188899
- [Background] Smith AD, Jull G, Schneider G, Frizzell B, Hooper RA, Sterling M. Cervical radiofrequency neurotomy reduces central hyperexcitability and improves neck movement in individuals with chronic whiplash. Pain Med. 2014 Jan;15(1):128-41. doi: 10.1111/pme.12262. Epub 2013 Oct 18. PMID 24138594
- [Background] Southerst D, Nordin MC, Cote P, Shearer HM, Varatharajan S, Yu H, Wong JJ, Sutton DA, Randhawa KA, van der Velde GM, Mior SA, Carroll LJ, Jacobs CL, Taylor-Vaisey AL. Is exercise effective for the management of neck pain and associated disorders or whiplash-associated disorders? A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Spine J. 2016 Dec;16(12):1503-1523. doi: 10.1016/j.spinee.2014.02.014. Epub 2014 Feb 15. PMID 24534390
- [Background] Stemper BD, Yoganandan N, Pintar FA. Validation of a head-neck computer model for whiplash simulation. Med Biol Eng Comput. 2004 May;42(3):333-8. doi: 10.1007/BF02344708. PMID 15191078
- [Background] Sterling M. A proposed new classification system for whiplash associated disorders--implications for assessment and management. Man Ther. 2004 May;9(2):60-70. doi: 10.1016/j.math.2004.01.006. PMID 15040964
- [Background] Sterling M. Differential development of sensory hypersensitivity and a measure of spinal cord hyperexcitability following whiplash injury. Pain. 2010 Sep;150(3):501-506. doi: 10.1016/j.pain.2010.06.003. Epub 2010 Jul 1. PMID 20594646
- [Background] Sterling M, Hendrikz J, Kenardy J. Compensation claim lodgement and health outcome developmental trajectories following whiplash injury: A prospective study. Pain. 2010 Jul;150(1):22-28. doi: 10.1016/j.pain.2010.02.013. Epub 2010 Mar 21. PMID 20307934
- [Background] Sterling M, Hendrikz J, Kenardy J. Similar factors predict disability and posttraumatic stress disorder trajectories after whiplash injury. Pain. 2011 Jun;152(6):1272-1278. doi: 10.1016/j.pain.2011.01.056. Epub 2011 Mar 10. PMID 21396780
- [Background] Sterling M, Hendrikz J, Kenardy J, Kristjansson E, Dumas JP, Niere K, Cote J, deSerres S, Rivest K, Jull G. Assessment and validation of prognostic models for poor functional recovery 12 months after whiplash injury: a multicentre inception cohort study. Pain. 2012 Aug;153(8):1727-1734. doi: 10.1016/j.pain.2012.05.004. Epub 2012 Jun 1. PMID 22658881
- [Background] Sterling M, Jull G, Kenardy J. Physical and psychological factors maintain long-term predictive capacity post-whiplash injury. Pain. 2006 May;122(1-2):102-8. doi: 10.1016/j.pain.2006.01.014. Epub 2006 Mar 9. PMID 16527397
- [Background] Sterling M, Jull G, Vicenzino B, Kenardy J, Darnell R. Physical and psychological factors predict outcome following whiplash injury. Pain. 2005 Mar;114(1-2):141-8. doi: 10.1016/j.pain.2004.12.005. Epub 2005 Jan 21. PMID 15733639
- [Background] Stewart MJ, Maher CG, Refshauge KM, Herbert RD, Bogduk N, Nicholas M. Randomized controlled trial of exercise for chronic whiplash-associated disorders. Pain. 2007 Mar;128(1-2):59-68. doi: 10.1016/j.pain.2006.08.030. Epub 2006 Oct 9. PMID 17029788
- [Background] Tate RL, Perdices M, Rosenkoetter U, Shadish W, Vohra S, Barlow DH, Horner R, Kazdin A, Kratochwill T, McDonald S, Sampson M, Shamseer L, Togher L, Albin R, Backman C, Douglas J, Evans JJ, Gast D, Manolov R, Mitchell G, Nickels L, Nikles J, Ownsworth T, Rose M, Schmid CH, Wilson B. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) 2016 Statement. Neuropsychol Rehabil. 2017 Jan;27(1):1-15. doi: 10.1080/09602011.2016.1190533. Epub 2016 Aug 8. PMID 27499422
- [Background] Teasell RW, McClure JA, Walton D, Pretty J, Salter K, Meyer M, Sequeira K, Death B. A research synthesis of therapeutic interventions for whiplash-associated disorder (WAD): part 2 - interventions for acute WAD. Pain Res Manag. 2010 Sep-Oct;15(5):295-304. doi: 10.1155/2010/640164. PMID 21038008
- [Background] Teasell RW, McClure JA, Walton D, Pretty J, Salter K, Meyer M, Sequeira K, Death B. A research synthesis of therapeutic interventions for whiplash-associated disorder (WAD): part 4 - noninvasive interventions for chronic WAD. Pain Res Manag. 2010 Sep-Oct;15(5):313-22. doi: 10.1155/2010/487279. PMID 21038010
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Winkelstein BA, Santos DG. An intact facet capsular ligament modulates behavioral sensitivity and spinal glial activation produced by cervical facet joint tension. Spine (Phila Pa 1976). 2008 Apr 15;33(8):856-62. doi: 10.1097/BRS.0b013e31816b4710. PMID 18404104
- [Background] Wu J, Zhou J, Liu C, Zhang J, Xiong W, Lv Y, Liu R, Wang R, Du Z, Zhang G, Liu Q. A Prospective Study Comparing Platelet-Rich Plasma and Local Anesthetic (LA)/Corticosteroid in Intra-Articular Injection for the Treatment of Lumbar Facet Joint Syndrome. Pain Pract. 2017 Sep;17(7):914-924. doi: 10.1111/papr.12544. Epub 2017 Feb 22. PMID 27989008
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Lord SM, Barnsley L, Bogduk N. Percutaneous radiofrequency neurotomy in the treatment of cervical zygapophysial joint pain: a caution. Neurosurgery. 1995 Apr;36(4):732-9. doi: 10.1227/00006123-199504000-00014. PMID 7596504
- [Background] Lovibond, S., & Lovibond, P. (1995). Manual for the Depression Anxiety Stress Scales (2nd ed.). Sydney: Psychology Foundation.
- [Background] Nikles, J. (2015). What are N-of-1 Trials? In J. Nikles & G. Mitchell (Eds.), The Essential Guide to N-of-1 Trials in Health (pp. 9-17). Dordrecht: Springer Netherlands.
- [Background] Parker, R. I., Vannest, K. J., & Brown, L. (2009). The improvement rate difference for single case research. Exceptional Children, 75, 135-150
- [Background] Podd D. Platelet-rich plasma therapy: origins and applications investigated. JAAPA. 2012 Jun;25(6):44-9. doi: 10.1097/01720610-201206000-00009. No abstract available. PMID 22693884
- [Background] SIRA - Guidelines for the management of acute whiplash associated disorders - for health professionals. (2014).
- [Background] Sullivan, M., Bishop, S., & Pivik, J. (1995). The pain catastrophizing scale: development and validation. Psychol Assess, 7, 524-532
- [Background] Van den Noortgate, W., & Onghena, P. (2007). The aggregation of single-case results using hierarchical linear models. The Behavior Analyst Today, 8(2), 196-209
- [Background] TRACsa - Clinical guidelines for best practice management of acute and chronic whiplash-associated disorders (2008).
- [Background] Jull, G., Sterling, M., Falla, D., et al. (2008). Whiplash, Headache and Neck Pain (1 ed.): Churchill Livingstone.
- See also: Oxford Centre for Evidence-Based Medicine Levels of Evidence Working Group(2011). The Oxford 2011 Levels of Evidence Table (Introduction) — http://www.cebm.net/index.aspx?o=5653